CLINICAL TRIAL: NCT06958588
Title: Pulsed Electromagnetic Field Therapy (PEMF) Compared to Conventional Mechanical Prophylaxis for Venous Thromboembolism Prophylaxis in Patients in the Intensive Care Unit (ICU)
Brief Title: Pulsed Electromagnetic Field Therapy or Pneumatic Compression VTE Prophylaxis
Acronym: SOPHIE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Science Valley Research Institute (Other)
Collaborators: Hospital Vera Cruz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAAE: 86295325.3.1001.0229
Record Dates: First submitted 2025-03-07; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-03

CONDITIONS: Venous Thromboembolism (VTE); Intensive Care Medicine; Venous Thromboembolism
Keywords: venous thromboembolism; Mechanical prophylaxis; Pulsed Electromagnetic Field Therapy (PEMF); ICU; intensive care unit
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperslim (Experimental): Pulsed Electromagnetic Field Therapy (PEMF)
  Interventions: Device: Experimental: Hyperslim
- Mechanical compression (Active Comparator): Intermittent pneumatic compression ( Covidien Kendall SCD 700®, Cardinal Health or Doctor Life 2600® Venosan)
  Interventions: Device: Active Comparator #1

INTERVENTIONS:
Device: Experimental: Hyperslim — The PEMF will be carried out using the Hyperslim® device. The Hyperslim® device is produced by Medical San (Lageado, RS, Brazil).
  Arms: Hyperslim
Device: Active Comparator #1 — The intermittent pneumatic compression group will use the devices Covidien Kendall SCD 700® (Cardinal Health) or Doctor Life 2600® (Venosan).
  Arms: Mechanical compression

SUMMARY:
Venous thromboembolism (VTE) is frequent in patients in the intensive care unit (ICU). Pharmacologic prophylaxis is sometimes contraindicated, and mechanical prophylaxis is used. The primary objective of the study is to compare Pulsed Electromagnetic Field Therapy (PEMF) with conventional mechanical prophylaxis for the prevention of VTE in patients in the ICU.

DETAILED DESCRIPTION:
This study is a prospective, randomized, open-label, active-controlled study, patients with indication for mechanical VTE prophylaxis or combined mechanical and pharmacological in the ICU from 2 selected sites in Brazil (Vera Cruz Hospital and Felicio Rocho Hospital, both in Belo Horizonte-MG, Brazil) will be enrolled after signing informed consent. All data will be recorded with a pre-established clinical recording file (CRF - RedCap) to demographics, risk factors, and clinical aspects of the patient's comorbidities.

A trained team member will perform clinical diagnosis and standard clinical evaluations, including imaging when indicated. Patients will be considered eligible if they are> 18 years old, have a PADUA score > 4 (medical patients) and/or Caprini > of 3 (surgical patients), and have a contraindication to pharmacological prophylaxis or indication to combined (pharmacological and mechanical VTE prophylaxis).

After signing informed consent, the patients will be screened and included in the study. After ICU admission, the patient will be interviewed by study investigators or trained physicians or nurses; inclusion patients will be randomized to receive either PEMF or intermittent pneumatic compression.

The devices will be placed in the ICUs following institutional standards and operational procedures. After randomization, trained physiotherapy and nurse teams will place and monitor each device. The intermittent pneumatic compression group will use the devices Covidien Kendall SCD 700® (Cardinal Health) or Doctor Life 2600® (Venosan). This group will have the device placed in the lower limbs, following the manufacturer's instructions, and monitored for 24 hours according to previous institutional protocol. This device will be kept full-time working in the patients while in the ICU.

The PEMF will be carried out using the Hyperslim® device. The Hyperslim® device is produced by Medical San (Lageado, RS, Brazil). It generates electromagnetic pulses through its pads, leading to local muscular supra-maximal contractions sustained for several seconds, increasing stress and workload without muscular adaptation. Its pads will be placed in the patient's lower limbs and used for 30 minutes thrice daily.

The critical care team will monitor patients 24 hours/day for VTE signs and symptoms, laboratory changes, and adverse local effects caused by machines like skin lesions, burns, and edema. A tolerability scale will be applied to every awake patient able to answer using a scale: 1= well tolerated; 2= tolerate with little discomfort; 3= tolerate with discomfort; 4= Not tolerated.

At the end of mechanical prophylaxis, patients will be evaluated for thromboembolic events, including diagnosis by imaging, with a mandatory Doppler ultrasound of the lower limbs at ICU discharge and 30 days post-randomization.

The primary efficacy outcome is a combination of symptomatic + asymptomatic VTE events at day 30 post randomization.

Evaluation also includes major bleeding events, defined as leading to transfusion of 2 or more units of blood or packed red cells, decrease in hemoglobin of 2 g/dL, bleeding in critical sites, defined as spinal, epidural, intraocular, intracranial, pericardial or retroperitoneal, local adverse events, including adverse events related to the use of the devices.

For descriptive statistics, mean and SD will be calculated for data following a Gaussian distribution.

The difference in VTE events between the two groups at the end of mechanical prophylaxis and day 30 will be tested using the intention-to-treat principle.

The efficacy analysis tests will be one-sided, with a type I error rate of 2·5%, assuming a two-sided 95% CI. The cumulative incidence of the composite events will be compared between the test and control groups, and the relative risk (RR) or risk ratio will be estimated. For the safety analysis, statistical tests will be two-sided, with a type I error rate of 5% and a two-sided 95% CI.

Tolerability, security, and facility to implement PEMF will be compared with intermittent pneumatic compression using an unpaired t-test.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years old in ICU
2. PADUA score> 4 (medical patients) and/or Caprini score> 3 (surgical patients)
3. Contraindication to pharmacological prophylaxis or indication to combined (pharmacological and mechanical VTE prophylaxis)

Exclusion Criteria:

1. Patients < 18 years old in ICU
2. Unable to use mechanical prophylaxis due to trauma, burns, fracture, or problems in inferior members that prevent the use of mechanical prophylaxis
3. Life expectations less than 24 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy outcome | 30 days
  The primary outcome is a composite of symptomatic and asymptomatic VTE (detected by mandatory Doppler ultrasound 24-48 hours after the end of mechanical prophylaxis or PEMF and on day 30 post-randomization) and death due to pulmonary embolism.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Ramacciotti, MD, Ph.D., Study Chair — Science Valley Research Organization
Locations (1):
- Hospital Vera Cruz, Belo Horizonte, MG, Brazil, Belo Horizonte, BH, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data can be made available upon requests directed to the corresponding author. Proposals will be reviewed based on scientific merit. After approval of a proposal, data can be shared through a secure online platform after signing a data access agreement.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: March 2025 to March 2030
Access Criteria: Anonymized participant data can be made available upon requests directed to the corresponding author. Proposals will be reviewed based on scientific merit. After approval of a proposal, data can be shared through a secure online platform after signing a data access agreement.

REFERENCES:
- [Background] Caprini JA. Mechanical methods for thrombosis prophylaxis. Clin Appl Thromb Hemost. 2010 Dec;16(6):668-73. doi: 10.1177/1076029609348645. Epub 2009 Oct 22. PMID 19850588
- [Background] Nicolaides AN, Fareed J, Spyropoulos AC, Kakkar RHL, Antignani PL, Avgerinos E, Baekgaard N, Barber E, Bush RL, Caprini JA, Clarke-Pearson DL, VAN Dreden P, Elalami I, Gerotziafas G, Gibbs H, Goldhaber S, Kakkos S, Lefkou E, Labropoulos N, Lopes RD, Mansilha A, Papageorgiou C, Prandoni P, Ramacciotti E, Rognoni C, Urbanek T, Walenga JM. Prevention and management of venous thromboembolism. International Consensus Statement. Guidelines according to scientific evidence. Int Angiol. 2024 Feb;43(1):1-222. doi: 10.23736/S0392-9590.23.05177-5. No abstract available. PMID 38421381
- [Background] Bounes F, Ferrandis R, Frere C, Helms J, Llau JV. European guidelines on peri-operative venous thromboembolism prophylaxis: first update.: Chapter 4: Prophylaxis in critical care patients. Eur J Anaesthesiol. 2024 Aug 1;41(8):582-588. doi: 10.1097/EJA.0000000000002011. Epub 2024 Jul 10. No abstract available. PMID 38957023
- [Background] Kearon C, Akl EA, Comerota AJ, Prandoni P, Bounameaux H, Goldhaber SZ, Nelson ME, Wells PS, Gould MK, Dentali F, Crowther M, Kahn SR. Antithrombotic therapy for VTE disease: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e419S-e496S. doi: 10.1378/chest.11-2301. PMID 22315268
- [Background] Schunemann HJ, Cushman M, Burnett AE, Kahn SR, Beyer-Westendorf J, Spencer FA, Rezende SM, Zakai NA, Bauer KA, Dentali F, Lansing J, Balduzzi S, Darzi A, Morgano GP, Neumann I, Nieuwlaat R, Yepes-Nunez JJ, Zhang Y, Wiercioch W. American Society of Hematology 2018 guidelines for management of venous thromboembolism: prophylaxis for hospitalized and nonhospitalized medical patients. Blood Adv. 2018 Nov 27;2(22):3198-3225. doi: 10.1182/bloodadvances.2018022954. PMID 30482763
- [Background] Ho KM, Chavan S, Pilcher D. Omission of early thromboprophylaxis and mortality in critically ill patients: a multicenter registry study. Chest. 2011 Dec;140(6):1436-46. doi: 10.1378/chest.11-1444. Epub 2011 Sep 22. PMID 21940768
- [Background] Fernando SM, Tran A, Cheng W, Sadeghirad B, Arabi YM, Cook DJ, Moller MH, Mehta S, Fowler RA, Burns KEA, Wells PS, Carrier M, Crowther MA, Scales DC, English SW, Kyeremanteng K, Kanji S, Kho ME, Rochwerg B. VTE Prophylaxis in Critically Ill Adults: A Systematic Review and Network Meta-analysis. Chest. 2022 Feb;161(2):418-428. doi: 10.1016/j.chest.2021.08.050. Epub 2021 Aug 19. PMID 34419428
- [Background] Lauzier F, Muscedere J, Deland E, Kutsogiannis DJ, Jacka M, Heels-Ansdell D, Crowther M, Cartin-Ceba R, Cox MJ, Zytaruk N, Foster D, Sinuff T, Clarke F, Thompson P, Hanna S, Cook D; Co-operative Network of Critical Care Knowledge Translation for Thromboprophylaxis (CONECCKT-T) Investigators; Canadian Critical Care Trials Group. Thromboprophylaxis patterns and determinants in critically ill patients: a multicenter audit. Crit Care. 2014 Apr 25;18(2):R82. doi: 10.1186/cc13844. PMID 24766968